CLINICAL TRIAL: NCT00341237
Title: Personalized Environment and Genes Study
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040053; 04-E-0053
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-11-25

CONDITIONS: Diabetes; Heart Disease; Asthma
Keywords: Genotype; Phenotype; Environmental Factor; Single Nucleotide Polymorphism; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- polymorphisms: Specimens are available to investigators in coded form to anonymously screen for the presence of single-nucleotide polymorphisms (SNPs) and other mutations in DNA.

SUMMARY:
Despite the overwhelming focus on genetic and genomic causes of human disease over the past two decades, it has been estimated that genetics is currently known to explain only 20% and 40% of the etiology of common disease. Thus, it is becoming increasingly apparent that human disease is a consequence of both genetic susceptibility and environmental exposures. Importantly, while individuals cannot change their genetic composition, we do have the ability both personally and as a society, to influence our environment, promoting health and decreasing the risk of disease. The Personalized Environment and Genes Study (PEGS) aims to determine how the environment and gene-environment interactions can inform our understanding of human health and disease. As science has evolved, so too has the science of this project. This evolution was reflected in a change in the title of this project from the Environmental Polymorphisms Registry (EPR) to the Personalized Environment and Genes Study (PEGS) to more accurately reflect the science that can be conducted. PEGS is a unique resource because of the depth of environmental phenotyping which includes extensive information from exposome surveys, as well as whole genome sequencing on a significant number of participants in the cohort. While it is small relative to genomic cohorts, none of these have the extensive environmental data that is present in PEGS. In addition, other cohorts with deep environmental data lack the depth of genomic data that is present in PEGS. Importantly, PEGS has already provided important analytic advances that are of great interest to and can be confirmed in larger cohorts such as All of Us.

The Personalized Environment and Genes Study (PEGS) aims to provide a resource for environmental health translational research by examining gene-environment interactions in health and disease. PEGS is an extension of two previous efforts where it began as a pilot study, the Environmental Polymorphisms Study (EPS; IRB# 02E9004) and was approved subsequently as a full protocol titled the Environmental Polymorphisms Registry (EPR) (IRB #04-E-N0053 and transitioned to its current ID# 04-E-0053). The EPR was envisioned as a phenotype-by-genotype registry of participants who had donated DNA samples, and who had agreed to be contacted for follow-up clinical translational studies based on their DNA genotypes. At the time, the only information available was a participant s age, sex, race, and ethnicity. Further phenotyping of a participant and/or any biospecimens obtained were investigated during a follow-up translational clinical study on participants recruited based on their genotype (hence phenotype-by-genotype) and the PEGS was the first recruit-by- genotype study at the NIH. Following a period focused on recruiting approximately 15,000 participants to enable genotyping of rare (approximately 1% minor allele frequency) single nucleotide polymorphisms (SNPs), the PEGS Consortium Project was undertaken in 2010- 2011 to examine, using the DNA of nearly 4,000 participants, approximately 700 SNPs in approximately 80 environmental response genes that work in concert with environmental exposures to elicit a phenotype. Several clinical follow-up studies, genotype-phenotype association studies, and publications have resulted from the PEGS Consortium Project.

To expand phenotype information available to researchers, the Health and Exposure Questionnaire was administered between 2013-2014. In 2017, a more detailed Exposome Questionnaire which includes questions relating to the external and internal exposome was administered. This was an important resource through which to integrate exposures with genotype-phenotype association studies.

Whole genome sequencing has now been performed on approximately 4700 participants who were reconsented for this purpose, as indicated above. Questionnaire data was fully adjudicated and combined in a robust and searchable database. With the increased power of the data available, the project was renamed as the Personalized Environment and Genes Study (PEGS) and rolled out in Sept. 2021.

DETAILED DESCRIPTION:
Study Description: The Personalized Environment and Genes Study (PEGS) integrates genetic and environmental data to understand disease etiology, identify disease risk factors, and improve disease prevention.

Objectives: The objective of PEGS is to provide a resource for environmental health translational research by examining environment and gene-environment interactions in health and disease. PEGS will incorporate exposure and health information with or without genomic information to address the following objectives.

* Primary Objective: To uncover novel environmental risk factors for the most prevalent health conditions and diseases.
* Secondary Objective: To use an environmental precision medicine framework to uncover genetic susceptibilities to specific environmental exposures that can ultimately be used to provide a fuller understanding of individual risks for diseases.

Endpoints:

Primary Endpoints:

1. Dichotomous phenotype (multiple analyses; each analysis is focused on a single dichotomous phenotype of clinical interest,

   or a group of mechanistically related dichotomous phenotypes) Example: asthma;
2. Continuous phenotype (multiple analyses; each analysis is focused on a clinically relevant continuous phenotype). Example: FEV1, an indicator of asthma severity.

Secondary Endpoints:

1. Phenome (simultaneous assessment of all clinically relevant phenotypes);
2. Exposome.

ELIGIBILITY:
* INCLUSION CRITERIA

In order to be eligible for participation in this study, an individual must meet all of the following criteria:

* Adults greater than or equal to 18 years of age
* If female, must not be (self-reported as) pregnant. At the time of enrollment, a pregnancy test will only be done at the PI s discretion.
* Able to understand and provide written informed consent
* Able to come to the NIEHS Clinical Research Unit (CRU) for enrollment and study-related visits/procedures.

EXCLUSION CRITERIA

An individual who does not meet the inclusion criteria listed above is excluded from participation in this study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sample from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2010-05-26 (Actual)

PRIMARY OUTCOMES:
Disease | End of study
  Genetic changes and disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Kirschner, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Personal information will be shared with researchers only if they meet one of three requirements: 1) an IRB-approved study protocol has approval from the PEGS Internal Advisory Committee or PEGS PI (NIEHS investigators only); or 2) have an IRB-approved study protocol listed in Apex. C as of 11/20/20; or 3) have obtained IRB approval for a new protocol. Demographic information will be shared with IRB-approved researchers conducting genotyping, exposure, or disease-specific callback studies, and this data is labeled only with PEGS PINs. Pediatric participants data is available to researchers under PEGS policies. DNA samples shared with researchers is labeled only with the PEGS PIN. Those who consent to whole genome/whole exome sequencing, their de-identified data is shared with NIH data repositories. Researchers with an IRB-approved study can access PEGS participant data through the repositories, however personally identifiable information (PII) is not stored in the repository.

REFERENCES:
- [Derived] Mack JA, Burkholder A, Akhtari FS, House JS, Sovio U, Smith GCS, Schmitt CP, Fargo DC, Hall JE, Motsinger-Reif AA. A multi-ancestry genome-wide association study identifies novel candidate loci in the RARB gene associated with hypertensive disorders of pregnancy. HGG Adv. 2025 Jan 9;6(1):100385. doi: 10.1016/j.xhgg.2024.100385. Epub 2024 Nov 22. PMID 39580622
- [Derived] Hussain S, Johnson CG, Sciurba J, Meng X, Stober VP, Liu C, Cyphert-Daly JM, Bulek K, Qian W, Solis A, Sakamachi Y, Trempus CS, Aloor JJ, Gowdy KM, Foster WM, Hollingsworth JW, Tighe RM, Li X, Fessler MB, Garantziotis S. TLR5 participates in the TLR4 receptor complex and promotes MyD88-dependent signaling in environmental lung injury. Elife. 2020 Jan 28;9:e50458. doi: 10.7554/eLife.50458. PMID 31989925
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-E-0053.html